CLINICAL TRIAL: NCT05249166
Title: Feeding for Accesible, Affordable and Healthy Childhood
Acronym: ALINFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Universidad Pública de Navarra (Other); Gobierno de Navarra (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ALINFA
Record Dates: First submitted 2021-12-09; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-01

CONDITIONS: Healthy Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Subjects assigned to this arm will follow the habitual recommendations to develop skills for a healthy diet. No specific foods or cooking methods will be applied
  Interventions: Other: Control
- ALINFA group (Experimental): This group will receive, in addition to the usual recommendations, meals, and foods designed to increase the healthiness of the diet. Foods and meals have been designed to increase the fiber content, decrease sugars and saturated fats, and limit salt intake.
  Interventions: Other: ALINFA

INTERVENTIONS:
Other: ALINFA — Comparing the usual recommendations with the healthy diet designed and developed
  Arms: ALINFA group
Other: Control — control group
  Arms: Control group

SUMMARY:
The main objective of this study was to evaluate the effectiveness of implementing a healthy eating vs traditional recommendations on the Medkid index of children in primary school. To do so, different companies involved in ALINFA project developed with the assessment of UNAV, CNTA and UPNA, a healthy bi-weekly menu.

ELIGIBILITY:
Inclusion Criteria:

* Adequate cultural level and comprehension of the clinical study from the legal tutors.
* To agree in taking part of the study.

Exclusion Criteria:

* Children presenting clinically relevant gastrointestinal malfunctions or structural anomalies, such as ulcers, chronic inflammatory diseases, etc. Even if they do not follow any pharmacological treatment at the moment of inclusion.
* Children with uncontrolled endocrine disorders.
* Children with any type of tumor/cancer within the last 5 years, or in current treatment.
* Children with any alimentary allergy.
* Children presenting any type of cognitive or psychic disorder
* Parents or legal tutors in which their future collaboration may not be the required, seen from the researchers' point of view.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Dietary Pattern (questionnaire) | Baseline
  Evaluate differences in dietary pattern between groups
Dietary pattern (questionnaire) | 8 week
  Evaluate differences in dietary pattern between groups
Dietary pattern (questionnaire) | Baseline vs 8 week
  Evaluated changes in dietary pattern

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Navas Carretero, PhD, Principal Investigator — University of Navarra
Locations (1):
- Center for Nutrition Research. University of Navarra, Pamplona, Navarre, Spain